CLINICAL TRIAL: NCT06746818
Title: Resilience Building Among Older Adults: the Heart Math Based Interventions for Posttraumatic Stress Disorder, Spirituality and Psychosocial Well-being
Acronym: Resilience
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Hashem El-Monshed, Associate Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EHEART
Record Dates: First submitted 2024-12-07; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
Keywords: Resilience; older adults; posttraumatic stress disorder; spirituality; psychosocial well-being
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The Heart Math Institute has been researching the relationship between the heart, brain, and body and its association to personal well-being and optimal functioning. Based on extensive research, the institute has developed a program that teaches participants the science behind and techniques designed to reduce the negative effects of stress and increase resilience (HeartMath Institute, 2020). The HeartMath intervention was conducted after the researcher successfully completed 13 hours (over two months) training of professional development in "The Resilience Heart TM: Trauma- Sensitive HeartMath Course" from HeartMath Institute.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): No care
- Intervention (Experimental): . The key components of Heart Math interventions include:
  1. Heart Rate Variability (HRV) Training: This involves biofeedback techniques to help individuals learn how to control their heart rate and promote emotional balance.
  2. Quick Coherence Technique: Participants are guided through a series of steps to shift their emotional state from stress to calmness, facilitating a sense of peace and emotional clarity.
  3. Focus on Positive Emotions: Encouraging individuals to cultivate feelings like gratitude and compassion can enhance resilience and overall mental well-being.
  4. Mindfulness Practices: Incorporating mindfulness helps individuals become more aware of their thoughts and feelings, allowing them to respond to stressors more effectively.
  Interventions: Behavioral: Heart Math interventions

INTERVENTIONS:
Behavioral: Heart Math interventions — . The key components of Heart Math interventions include:
  1. Heart Rate Variability (HRV) Training: This involves biofeedback techniques to help individuals learn how to control their heart rate and promote emotional balance.
  2. Quick Coherence Technique: Participants are guided through a series of steps to shift their emotional state from stress to calmness, facilitating a sense of peace and emotional clarity.
  3. Focus on Positive Emotions: Encouraging individuals to cultivate feelings like gratitude and compassion can enhance resilience and overall mental well-being.
  4. Mindfulness Practices: Incorporating mindfulness helps individuals become more aware of their thoughts and feelings, allowing them to respond to stressors more effectively.
  Arms: Intervention

SUMMARY:
Resilience building among older adults: The Heart Math based interventions for posttraumatic stress disorder, spirituality and psychosocial well-being.

Resilience building among older adults is critically important, especially in the context of mental health challenges such as posttraumatic stress disorder (PTSD). Interventions that promote well-being through innovative methods can significantly enhance the quality of life in this demographic. One such approach is the Heart Math-based intervention, which integrates techniques for emotional regulation, stress reduction, and overall psychosocial well-being.

Understanding Heart Math Interventions The HeartMath training program, developed by the HeartMath Institute, focuses on teaching individuals self-regulation skills that promote heart-brain coherence. This state of coherence has been associated with improved cognitive function, emotional stability, and physical health. By integrating this training into the care of older adults with PTSD, nurses can play a pivotal role in addressing the complex emotional and psychological needs of this population.

. The key components of Heart Math interventions include:

1. Heart Rate Variability (HRV) Training: This involves biofeedback techniques to help individuals learn how to control their heart rate and promote emotional balance.
2. Quick Coherence Technique: Participants are guided through a series of steps to shift their emotional state from stress to calmness, facilitating a sense of peace and emotional clarity.
3. Focus on Positive Emotions: Encouraging individuals to cultivate feelings like gratitude and compassion can enhance resilience and overall mental well-being.
4. Mindfulness Practices: Incorporating mindfulness helps individuals become more aware of their thoughts and feelings, allowing them to respond to stressors more effectively.

Impact on PTSD and Psychosocial Well-Being

For older adults experiencing PTSD, Heart Math interventions can offer several benefits:

* Reduced Anxiety and Stress: By learning techniques to control physiological responses to stress, older adults can experience lower levels of anxiety and an improved ability to manage PTSD symptoms.
* Enhanced Emotional Regulation: These interventions help individuals to better regulate their emotions, reducing instances of emotional dysregulation often seen in PTSD.
* Greater Spiritual Connection: Engaging in practices that promote positive emotions and mindfulness can enhance a sense of spirituality and purpose, which is particularly beneficial in aging populations.
* Improved Social Support: Group-based Heart Math interventions can foster social connections, which play a key role in building resilience among older adults.
* Overall Well-Being: Focusing on emotional health fosters a holistic outlook, improving physical, mental, and spiritual well-being.

Practical Implementation

1. Workshops and Group Sessions: Facilitate group workshops that incorporate Heart Math techniques. This encourages peer support and sharing of experiences.
2. Personal Coaching: Offer one-on-one sessions to guide older adults through Heart Math practices, tailored to their specific needs and trauma experiences.
3. Follow-Up and Support: Establish ongoing support systems, such as regular check-ins or additional resources, to help maintain the benefits gained through the interventions.
4. Integrate into Existing Programs: Consider incorporating these techniques into existing mental health programs targeting older adults, enhancing current offerings with a focus on resilience.

summary Heart Math-based interventions present a promising approach to resilience building among older adults, particularly those dealing with PTSD. By addressing emotional regulation, enhancing spiritual well-being, and fostering psychosocial support, these interventions can lead to significant improvements in quality of life and mental health outcomes. As the population of older adults continues to grow, such innovative approaches will be essential in supporting their mental health and emotional resilience.

Research hypothesis: Older adults with PTSD who participate in HeartMath training program will show a statistically significant increase in resilience, spiritualty, and psychosocial wellbeing compared to those who do not participate in the program Setting: Elderly homes, Damanhour city, Elbehaira Governorate, Egypt. Subject: 120 older adults with PTSD. Tools: The posttraumatic Diagnostic scale, The Connor Davidson Resilience scale-10, Spiritual wellbeing scale, and psychosocial wellbeing questionnaire.

ELIGIBILITY:
Inclusion Criteria:

- Older adults aged 60 or more for both the control and study groups.

Exclusion Criteria:

* NA

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Tool II: The Posttraumatic Diagnostic Scale (The PDS-5) | through study completion, an average of 1 year
  Primary Outcome Measure: The PDS-5 is a self-report instrument that involves 24 elements and evaluates PTSD symptom severity in the past month in accordance with DSM-5 criteria (Foa et al., 2016). The PDS-5 begins with trauma-history screen questions to assess the trauma history of the participant. Twenty questions were devised to assess the presence and severity of the PTSD symptoms in relation to the index trauma; symptom questions were based on the DSM-5 symptom clusters of intrusion (Items 1-5), avoidance (Items 6 -7), changes in mood and cognition (Items 8 -14), and arousal and hyper-reactivity (Items 15-20).

SECONDARY OUTCOMES:
Tool III: The Connor-Davidson Resilience Scale-10-Item | through study completion, an average of 1 year
  The original Connor-Davidson Resilience Scale 10 (CDRISC 10) was developed by Campbell-Sills & Stein (2007) that was prepared based on the CD-RISC 25 (Connor & Davidson, 2003) comprises 10 self-report items, each rated on a Likert-type scale from 0 (not true at all) to 4 (true nearly all the time). In its original version, all of the 10 items load on a single dimension. The respondents complete the scale based on the degree to which they admit each item on the scale was applicable to them in the preceding 1 month. The total score could range from 0 to 40 with higher scores indicating greater resilience of the respondent.
Tool IV: Spiritual Well-being Scale | through study completion, an average of 1 year
  This scale was developed by Ellison (1983). It was widely used and well validated scale (Ellison & Smith, 1991). It is designed to assess religious and existential well-being. It was translated into Arabic language by Musa & Pevalin (2012) and proved to be valid. The scale comprises 20 statements. It is consisting of two subscales of 10 items each. The Religious Well-Being (RWB) subscale assesses the degree to which individuals report that they experience a satisfying relationship with God. Items of the Existential Well-Being (EWB) subscale relate to a sense of life satisfaction and purpose. Negatively worded items are reverse scored. Even numbered items assess existential well-being and odd numbered items assess religious well-being. The responses are rated on a 6-point Likert scale ranging from (1) indicating "strongly disagree" to (6) indicating "strongly agree".
Tool V: Psychosocial Wellbeing Questionnaire | through study completion, an average of 1 year
  It was developed by HalimahAwang et al., (2021) , which composed of 17 statements, eight positive and nine negative related to the outlook on life as experienced by the respondents in the past six months. It covering the domains of psychosocial wellbeing which include loneliness, life satisfaction and happiness. Each statement was measured on a five-point Likert scale where 1=never, 2=rarely, 3=sometimes, 4=often and 5=always.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura U, Al Mansurah, Egypt